CLINICAL TRIAL: NCT03403439
Title: Relative Bioavailability of a Single Oral Dose of BI 1015550 When Administered Alone or in Combination With Multiple Oral Doses of Itraconazole in Healthy Male Subjects
Brief Title: This Study in Healthy Men Tests How Itraconazole Influences the Amount of BI 1015550 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0015; 2017-003452-23 (EudraCT Number)
Record Dates: First submitted 2018-01-12; First posted 2018-01-18 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 1015550 alone (R) / itraconazole + BI 1015550 (T) (Experimental): Participants were administered single dose of BI 1015550 6 milligram (mg) tablet orally with 240 milliLitre (mL) of water after an overnight fast of at least 10 hours on Day 1 of Visit 2. Again participants were administered itraconazole plus BI 1015550; participants received 12 days of itraconazole treatment (200 mg itraconazole solution given orally once daily with 240 mL of water after an overnight fast of at least 9 h) from Day -3 to Day 9 of Visit 3 combined with a single dose of 6 mg BI 1015550 on the fourth day (Day 1) of the itraconazole treatment (1 hour after the itraconazole administration). The BI 1015550 single doses of treatments R and T were separated by a wash-out period of at least 10 days.
  Interventions: Drug: BI 1015550; Drug: itraconazole

INTERVENTIONS:
Drug: BI 1015550 — single dose of BI 1015550 6 milligram (mg) tablet orally with 240 milliLitre (mL) of water after an overnight fast of at least 10 hours
  Other Names: Nerandomilast; JASCAYD®
Drug: itraconazole — 200 mg itraconazole solution given orally once daily with 240 mL of water after an overnight fast of at least 9 h

SUMMARY:
The primary objective of this trial is to investigate whether and to what extent co-administration of multiple doses of itraconazole affect single dose pharmacokinetics of BI1015550, i.e. to compare the relative bioavailability of 6 mg BI 1015550 when given alone (reference, treatment R) to the relative bioavailability of 6 mg of BI 1015550 given on the 4th day of a 12-day-treatment with itraconazole (test, treatment T) following oral administration in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (BP (Blood Pressure), PR (Pulse Rate)), 12-lead ECG (Electrocardiogram), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP (Blood Pressure), PR (Pulse Rate) or ECG (Electrocardiogram)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm (beats per minute)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders, including but not limited to mood disorders and any history of suicidality.
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients or other Azoles )
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was as an open-label, fixed-sequence trial with 2 treatments, administered to healthy male participants to compare itraconazole + BI 1015550 (T) with BI 1015550 alone (R). The BI 1015550 single doses of treatments R and T were separated by a wash-out period of at least 10 days.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist site which would then ensure that they (all participants) met all inclusion/exclusion criteria. Participants were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Period: Treatment Period 1 + Washout (7 days)
Arm/Group | BI 1015550 alone (R) / itraconazole + BI 1015550 (T)
Started | 16
Completed | 16
Not Completed | 0
Period: Treatment Period 2 (21 days)
Arm/Group | BI 1015550 alone (R) / itraconazole + BI 1015550 (T)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all subjects who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Arm/Group | BI 1015550 Alone (R) / Itraconazole + BI 1015550 (T)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 to 119 Hours
Description: Area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 to 119 hours (h) (AUC0-119). Standard error is actually geometric standard error. Geometric mean (gMean) is actually adjusted geometric mean. Pharmacokinetic samples were collected at 3:00 hours:minutes (h:m) prior to drug administration and at 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00, 34:00, 47:00, 71:00, 95:00 and 119:00 h:m after drug administration during Visit 2 and Visit 3. Additionally at 143:00, 167:00, 191:00 and 215:00 h:m after drug administration during Visit 3.
Time Frame: Up to 215 hours (Please check measure description for detailed timeframe)
Population: Pharmacokinetic (PK) set (PKS):
  The PKS included all subjects from the TS who provided at least 1 primary or secondary PK parameter that was not excluded. Thus, a subject was included in the PKS, even if he contributed only 1 PK parameter value for 1 period to the statistical assessment.
Measure: Geometric Mean (Standard Error); unit: nanomole (nmol)*h/Litre (L)
Groups:
- itraconazole + BI 1015550 (T): Participants were administered itraconazole plus BI 1015550; 12 days of itraconazole treatment (200 mg itraconazole solution given orally once daily with 240 mL of water after an overnight fast of at least 9 h) from Day -3 to Day 9 of Visit 3 combined with a single oral dose of 6 mg BI 1015550 on the fourth day (Day 1) of the itraconazole treatment (1 hour after the itraconazole administration).
- BI 1015550 alone (R): Participants were administered alone with single dose of BI 1015550 6 mg tablet orally with 240 mL of water after an overnight fast of at least 10 hours on Day 1 of Visit 2.
Arm/Group | itraconazole + BI 1015550 (T) | BI 1015550 alone (R)
Number analyzed (Participants) | 16 | 16
nanomole (nmol)*h/Litre (L) | 2073.40 (NA) — Geometric standard error = 1.07 | 933.44 (NA) — Geometric standard error = 1.07
Statistical Analysis 1: Comparison: itraconazole + BI 1015550 (T) vs BI 1015550 alone (R); The analysis of variance (ANOVA) model included effects accounting for the following sources of variation: 'subject' and 'treatment'. The effect 'subject' was considered as random, whereas the effect 'treatment' was considered as fixed. No hypothesis was tested and no acceptance range was specified; Test type: Other; Geometric Mean (T/R) ratio (%) = 222.13, 90% CI 2-sided [203.47 to 242.49] — To get, gMean ratio (T/R) and confidence interval, least square estimates of log-transformed PK endpoint for T and R were back transformed to original scale. Intra-individual geometric coefficient of variance (%) = 14.2

2. Primary Outcome: Maximum Measured Concentration of the BI 1015550 in Plasma
Description: Maximum measured concentration of the BI 1015550 in plasma (Cmax). Standard error is actually geometric standard error. Geometric mean is actually adjusted geometric mean. Pharmacokinetic samples were collected at 3:00 h:m prior to drug administration and at 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00, 34:00, 47:00, 71:00, 95:00 and 119:00 h:m after drug administration during Visit 2 and Visit 3. Additionally at 143:00, 167:00, 191:00 and 215:00 h:m after drug administration during Visit 3.
Time Frame: Up to 215 hours (Please check measure description for detailed timeframe)
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol/L
Arm/Group | itraconazole + BI 1015550 (T) | BI 1015550 alone (R)
Number analyzed (Participants) | 16 | 16
nmol/L | 162.39 (NA) — Geometric standard error = 1.06 | 126.91 (NA) — Geometric standard error = 1.06
Statistical Analysis 1: Comparison: itraconazole + BI 1015550 (T) vs BI 1015550 alone (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean (T/R) ratio (%) = 127.96, 90% CI 2-sided [117.65 to 139.17] — To get, gMean ratio (T/R) and confidence interval, least square estimates of log-transformed PK endpoint for T and R were back transformed to original scale. Intra-individual geometric coefficient of variance (%) = 13.6

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf). Standard error is actually geometric standard error. Geometric mean is actually adjusted geometric mean. Pharmacokinetic samples were collected at 3:00 h:m prior to drug administration and at 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00, 34:00, 47:00, 71:00, 95:00 and 119:00 h:m after drug administration during Visit 2 and Visit 3. Additionally at 143:00, 167:00, 191:00 and 215:00 h:m after drug administration during Visit 3.
Time Frame: Up to 215 hours (Please check measure description for detailed timeframe)
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol*h/L
Arm/Group | itraconazole + BI 1015550 (T) | BI 1015550 alone (R)
Number analyzed (Participants) | 16 | 16
nmol*h/L | 2183.22 (NA) — Geometric standard error = 1.08 | 952.27 (NA) — Geometric standard error = 1.08
Statistical Analysis 1: Comparison: itraconazole + BI 1015550 (T) vs BI 1015550 alone (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean (T/R) ratio (%) = 229.26, 90% CI 2-sided [207.82 to 252.93] — To get, gMean ratio (T/R) and confidence interval, least square estimates of log-transformed PK endpoint for T and R were back transformed to original scale. Intra-individual geometric coefficient of variance (%) = 15.9

ADVERSE EVENTS:
Time Frame: From the first BI 1015550 administration until end of trial, up to 28 days (i.e. 7 days for BI 1015550, 3 days for itraconazole and up to 18 days for itraconazole + BI 1015550).
Description: TS
Groups:
- BI 1015550: Participants were administered single dose of BI 1015550 6 mg tablet orally with 240 mL of water, in treatment R.
- itraconazole: Participants were administered itraconazole 200 mg solution orally once daily with 240 mL of water after an overnight fast of at least 9 h, in treatment T only for 3 days from Day -3 to Day -1 of Visit 3.
- itraconazole + BI 1015550: Participants were administered itraconazole plus BI 1015550; participants received 9 days of itraconazole treatment (200 mg itraconazole solution given orally once daily with 240 mL of water after an overnight fast of at least 9 h) from Day 1 to Day 9 of Visit 3 combined with a single dose of 6 mg BI 1015550 on Day 1 (1 hour after the itraconazole administration).
Arm/Group | BI 1015550 | itraconazole | itraconazole + BI 1015550
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 5/16 | 5/16 | 9/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1015550 (N=16) | itraconazole (N=16) | itraconazole + BI 1015550 (N=16)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 5
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 2
Thirst (General disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03403439/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT03403439/SAP_001.pdf